CLINICAL TRIAL: NCT06742385
Title: Evaluation of a Remote Monitoring Application in the Follow-up of Patients With Active Inflammatory Bowel Diseases: The SECURITY Trial
Brief Title: Evaluation of a Remote Monitoring Application in the Follow-up of Patients With Active Inflammatory Bowel Diseases
Acronym: SECURITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: AbbVie (Industry); Semeia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GETAID-2023-02
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial comparing two strategies to following-up patients with active IBD; Active arm: alerts activated, Control arm: alerts disabled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): Both arms are equipped with the application, data are collected via the application and telemonitoring with alerts to the care team are activated in the active telemonitoring arm.
  Interventions: Device: MedicWise
- Control arm (No Intervention): Both arms are equipped with the application, data are collected via the application and telemonitoring with alerts to the care team are inactivated in the active control arm.

INTERVENTIONS:
Device: MedicWise — * Both arms are equipped with the application, data are collected via the application and telemonitoring with alerts to the care team are activated in the active telemonitoring arm.
  * Data are collected in both arms at baseline, M3, M6, M9 and M12
  * Each center defines who handles alerts internally (physicians, IBD nurses, others, etc.) according to its internal organization. The application does not impose an internal operation.
  * the alert thresholds are identical and fixed for all centers during the study. Within the framework of the study, alerts are defined according to the study's modalities but cannot be modified by the centers.
  * Participating sites will have no obligation to respond to alerts.
  * Randomization will be stratified by centers and by diseases (Crohn and UC) with unbalanced blocks of randomization
  Arms: Active arm

SUMMARY:
Telemonitoring is of definite theoretical interest for patients suffering from chronic diseases and could help to improve monitoring of treatment efficacy and tolerance, and hence remission and quality of life. Reimbursement is now planned in France for devices that have demonstrated a positive effect on patient intake. However, available studies testing different tools in IBD have shown no significant improvement in disease control or quality of life. Nevertheless, major secondary endpoints such as reduced hospitalization, complications and healthcare costs have been demonstrated. Several biases have been identified to explain these disappointing results, such as the heterogeneity of the tools/applications tested, methodological limitations concerning the main objective and technological limitations of the tools evaluated.

We propose here to evaluate the impact of a tight remote monitoring through digital tool on disease control, in patients with active IBD, thanks to the MedicWise platform. The technology of the MedicWise solution enables the automatic collection of a wide range of biological and healthcare consumption data, thus limiting the need for patient input. MedicWise has obtained the CE label and is already used and reimbursed in France in other chronic diseases. The SECURITY trial proposes to evaluate the impact of a tight remote monitoring through digital tool on time spent in remission. Improvement of IBD related disability is also a major secondary objective of the study. It also has the following secondary objectives to analyze the impact of this tool on the organization of care teams caring for patients with IBD.

DETAILED DESCRIPTION:
Telemonitoring is of definite theoretical interest for patients suffering from chronic diseases and could help to improve monitoring of treatment efficacy and tolerance, and hence remission and quality of life. Reimbursement is now planned in France for devices that have demonstrated a positive effect on patient intake. However, available studies testing different tools in IBD have shown no significant improvement in disease control or quality of life. Nevertheless, major secondary endpoints such as reduced hospitalization, complications and healthcare costs have been demonstrated. Several biases have been identified to explain these disappointing results, such as the heterogeneity of the tools/applications tested, methodological limitations concerning the main objective and technological limitations of the tools evaluated.

We propose here to evaluate the impact of a tight remote monitoring through digital tool on disease control, in patients with active IBD, thanks to the MedicWise platform. The technology of the MedicWise solution enables the automatic collection of a wide range of biological and healthcare consumption data, thus limiting the need for patient input. MedicWise has obtained the CE label and is already used and reimbursed in France in other chronic diseases. The SECURITY trial proposes to evaluate the impact of a tight remote monitoring through digital tool on time spent in remission. Improvement of IBD related disability is also a major secondary objective of the study. It also has the following secondary objectives to analyze the impact of this tool on the organization of care teams caring for patients with IBD.

Main objective: To evaluate whether tight control through remote monitoring device improves disease activity compare to standard of care in patients with active Inflammatory Bowel Disease (IBD).

ELIGIBILITY:
Inclusion Criteria:

* CD/UC patients with a validated diagnosis
* Patients age > 18 years
* IBD with clinical signs of PRO2 activity leading to modification of medical treatment: introduction of a new treatment, or change of dose or addition of a treatment (corticoids, ASA, IS, biotherapy (a 4 week induction phase is authorized
* Patients willing and able to participate in the collection of data via SEMEIA App on their smartphone
* Patients agreeing to participate for 12 months

Exclusion Criteria:

* Patients with an inability to use a smartphone and email
* Patients < 18 years old
* Digestive surgery expected within 3 months
* Pregnancy at baseline
* Patients with an history of sub-total colectomy, coloproctectomy, digestive ostomy, extensive or multiple intestinal resections with sequelae of diarrhoea, short bowel syndrome.
* Patients who have had recent digestive surgery (ileal resection < 6 months) Patients with any other uncontrolled somatic or psychiatric pathology
* Patients enrolled in a trial with an investigational treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-09-18 (Estimated); Study Completion 2028-09-18 (Estimated)

PRIMARY OUTCOMES:
Percentage of cumulative time spent in symptomatic remission within 12 months | 12 months
  Percentage of cumulative time spent in symptomatic remission within 12 months
  Time spent in symptomatic remission defined by (PRO2):
  MC: abdominal pain ≤ 1 and stool frequency ≤ 3 defined clinical remission in CD, both not worsening compared from inclusion
  UC: absence of rectal bleeding (score 0) and stool frequency score ≤ 1, both not worsening compared with inclusion

SECONDARY OUTCOMES:
Average value of IBD disk change from baseline over 12 months (M3, M6, M9 and M12) | 12 months
  Average value of IBD disk change from baseline over 12 months (M3, M6, M9 and M12)
Average value of IBD disk change from baseline over 12 months | 12 months
  Average value of IBD disk change from baseline over 12 months
Patient report outcomes (PR02), questionnaire to assess this outcome measure at M6 and M12 | 6 and 12 months
  Patient report outcomes (PR02), questionnaire to assess this outcome measure at M6 and M12
Short Inflammatory Bowel Disease (S-IBDQ) delta mean value between inclusion and M12 (The total score ranges from 10 to 70, with the higher the score, the better the quality of life.) | 12 months
  Short Inflammatory Bowel Disease (S-IBDQ) delta mean value between inclusion and M12
Average value of Short Inflammatory Bowel Disease (S-IBDQ) delta mean value between inclusion and M12 (The total score ranges from 10 to 70, with the higher the score, the better the quality of life.) change from baseline over 12 months | 12 months
  Average value of Short Inflammatory Bowel Disease (S-IBDQ) delta mean value between inclusion and M12 (The total score ranges from 10 to 70, with the higher the score, the better the quality of life.) change from baseline over 12 months
Number of contacts / consultations / hospitalizations during 12 months | 12 months
  Number of contacts / consultations / hospitalizations during 12 months
Medication and care compliance/consumption over 12 months | 12 months
  Medication and care compliance/consumption over 12 months
number of complications (AE/SAE, hospitalizations, surgeries) over 12 months | 12 months
  number of complications (AE/SAE, hospitalizations, surgeries) over 12 months
Satisfaction questionnaires (patients/care team) at M12 | 12 months
  Satisfaction questionnaires (patients/care team) at M12

CONTACTS AND LOCATIONS:
Locations (1):
- Institut des MICI, Neuilly-sur-Seine, France, France

IPD SHARING:
Plan to Share IPD: Undecided